CLINICAL TRIAL: NCT04514224
Title: Implementation of a Health Information Technology System for Young African American Women Into Community-Based Clinical Sites
Brief Title: Gabby Implementation: Parent Protocol
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: H-36816; 1R18HS025131-01 (AHRQ)
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Preconception Care
Keywords: Healthy Start program; Community Health Centers; Implementation Science Research; Uptake; Organizational Readiness; Health Information Technology; Embodied Conversational Agent; Preconception Health; Black and African American women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Healthy Start Program 1: Community Partner with HRSA-funded Healthy Start designation and services a patient population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Community Health Center 1: Community Partner with Community Health Center or Federally Qualified Community Health Center designation and services a client population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Healthy Start Program 2: Community Partner with HRSA-funded Healthy Start designation and services a patient population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Community Health Center 2: Community Partner with Community Health Center or Federally Qualified Community Health Center designation and services a client population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Healthy Start Program 3: Community Partner with HRSA-funded Healthy Start designation and services a patient population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Community Health Center 3: Community Partner with Community Health Center or Federally Qualified Community Health Center designation and services a client population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Healthy Start Program 4: Community Partner with HRSA-funded Healthy Start designation and services a patient population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Community Health Center 4: Community Partner with Community Health Center or Federally Qualified Community Health Center designation and services a client population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Healthy Start Program 5: Community Partner with HRSA-funded Healthy Start designation and services a patient population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation
- Healthy Start Program 6: Community Partner with HRSA-funded Healthy Start designation and services a patient population with over 50% identifying African American and/or Black
  Interventions: Other: Gabby implementation; Other: Evaluate the Gabby implementation

INTERVENTIONS:
Other: Gabby implementation — Iimplement an evidence-based preconception care intervention, Gabby, into community-based health settings
Other: Evaluate the Gabby implementation — Assess implementation outcomes using the Proctor Implementation Outcomes Framework

SUMMARY:
The Gabby Preconception Care program is an innovative communication system designed to identify and mitigate or resolve health risks for young Black and African American (AA) women before pregnancy, as a means of reducing racial health disparities in birth outcomes. The system uses embodied conversational agent technology the investigators call "Gabby," who empathically interacts with users to assess health risks and delivers interventions to resolve or mitigate these risks. This research team has been working on the "Gabby" Preconception Care program, which features Virtual Patient Advocate (VPA) technology, for over seven years and the system is now ready for dissemination beyond the research environment and into the clinical and community context. The purpose of this project is to examine the implementation and dissemination process of the evidence-based Gabby Program.

Caseworkers at Healthy Start (HS) Programs and healthcare providers at Community Health Centers (CHC's) do not have time to assess for the over 100 preconception health risks that can impact birth outcomes; our system can assist by streamlining that assessment to create a personalized list of risks.Gabby will be introduced/released to sites as part of their standard of care where patients and clients can then share their list with healthcare providers and case workers/managers to make their in-person interactions much more effective. Studies by the research team have shown that Gabby reduces health risks by 25 percent among young Black and AA women. The investigators will evaluate the success of the implementation process through both quantitative and qualitative measures including key informant telephone interviews and guidance from a Gabby Toolkit Advisory Board in order to prepare an implementation toolkit that can be used to facilitate broader dissemination. The Gabby program will not be evaluated as a research intervention, as this has been done previously, instead, how well the Gabby program worked within each site will be assessed.

DETAILED DESCRIPTION:
The investigators' implementation approach includes: 1) engaging 6 Healthy Starts and 4 CHCs and assessing the workflow and readiness of these clinical sites; 2) implementing the Gabby program for a period of 3-6 months at each of these clinical sites; 3) assembling a preliminary, revised, and final implementation toolkit; and 4) broadly disseminating the toolkit and results of the implementation. Input from a Gabby Toolkit Advisory Board will guide implementation efforts and toolkit development to be used for wider dissemination into other clinical based sites.

Data sources will include qualitative and quantitative methods, such as surveys/ assessments, key informant interviews, system-generated data, learning communities, and implementation logs. Evaluation will focus on site recruitment, training, and engagement; client engagement; clinical risk reduction; toolkit, technical assistance, and support resources; and dissemination efforts.

ELIGIBILITY:
Inclusion Criteria:

For staff at Healthy Start sites and Community Health Centers

* Staff (community health workers, social workers, clinicians, administrators) who work at a participating site
* Trained about the Gabby system by the investigators
* Speak and read English

For Gabby system users

* Women who identify as black or African American who are clients of a participating Healthy Start site or receive care at a participating Community Health Center
* Currently not pregnant
* Speaks and read English
* Has access to a smartphone or laptop/tablet
* Has internet access
* Plans to use the Gabby system for 6 months

Exclusion Criteria:

For Staff at Healthy Start sites and Community Health Centers

* None

For Gabby system users

* None

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of staff members at participating sites and clients who use the Gabby system. The staff will be from the 6 selected Healthy Start sites and the 6 selected Community Health Centers who volunteer to participate by responding to a survey, being interviewed, or participating in a focus group about implementation of the Gabby program. The clients will be adult eligible women who receive services from one of the participating sites who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Acceptability of Gabby system by staff | 6 months
  Information about the acceptability of the Gabby system will be gleaned form qualitative and quantitative data. Virtual interviewers of key staff will be done informed by an interview guide to collect the qualitative data. The quantitative data will be assessed using an investigator developed 33-question Likert scale-based survey. Responses along the 5-point Likert scale will consist of Strongly Disagree (1), Disagree (2), Neutral (3), Agree (4), Strongly Agree (5). Higher score from acceptability related questions indicate greater acceptability.
Feasibility of Gabby system by staff | 6 months
  Information about the feasibility of the Gabby system will be gleaned form qualitative and quantitative data. Virtual interviewers of key staff will be done informed by an interview guide to collect the qualitative data. The quantitative data will be assessed using an investigator developed 33-question Likert scale-based survey. Responses along the 5-point Likert scale will consist of Strongly Disagree (1), Disagree (2), Neutral (3), Agree (4), Strongly Agree (5). Higher score from feasibility related questions indicate greater feasibility.

SECONDARY OUTCOMES:
Total number of preconception health risks for Gabby users | 6 months
  The total number of preconception risks is collected during the client/patient's interaction with the Gabby system and will be obtained from Gabby system reports produced by the Gabby System server
Change in number of preconception risks at 3 months | baseline, 3 months
  The number of preconception risks is collected during the client/patient's interaction with the Gabby system and will be obtained from Gabby system reports produced by the Gabby System server
Change in number of preconception risks at 6 months | baseline, 6 months
  The number of preconception risks is collected during the client/patient's interaction with the Gabby system and will be obtained from Gabby system reports produced by the Gabby System server
Stage of change for each preconception risk identified | 6 months
  The client's stage of change for each preconception risk is collected during the client/patient's interaction with the Gabby system and will be obtained from Gabby system reports produced by the Gabby System server
Number of Gabby sessions by user | 6 months
  The Gabby system records the number of log-ons/sessions for each user which will be obtained from Gabby system reports produced by the Gabby System server.
Total number of minutes used Gabby | 6 months
  The Gabby system records the number of minutes of each session for every user which will be obtained from Gabby system reports produced by the Gabby System server.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jack, MD, Principal Investigator — Boston Medical Center, Family Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walter AW, Julce C, Sidduri N, Yinusa-Nyahkoon L, Howard J, Reichert M, Bickmore T, Jack BW. Study protocol for the implementation of the Gabby Preconception Care System - an evidence-based, health information technology intervention for Black and African American women. BMC Health Serv Res. 2020 Sep 21;20(1):889. doi: 10.1186/s12913-020-05726-0. PMID 32958031